CLINICAL TRIAL: NCT01207557
Title: A Randomized Controlled Trial of the Effectiveness of the Ottawa Influenza Decision Aid - A Component of the "Optimizing Healthcare Workers Interpandemic Vaccine Uptake in Acute and Long-term Care" CIHR Project
Brief Title: A Randomized Controlled Trial of the Effectiveness of the Ottawa Influenza Decision Aid
Acronym: OIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bruyère Health Research Institute. (Other); Providence Health & Services (Other); Canadian Center for Vaccinology (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TPA 90189
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Influenza
Keywords: Healthcare personnel; influenza; immunization; flu; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard education only (Active Comparator): 50% of non-immunized personnel 4 weeks following start of campaign will be given standard education materials and tested on their confidence with their immunization decision
  Interventions: Behavioral: Standard Education Only
- Standard Education plus OIDA (Active Comparator): 50% of non-immunized personnel 4 weeks following start of campaign will be given standard education materials plus the Ottawa Influenza Decision Aid and tested on their confidence with their immunization decision
  Interventions: Behavioral: Standard Education Plus OIDA

INTERVENTIONS:
Behavioral: Standard Education Only — 50% of non-immunized personnel 4 weeks following start of campaign will be given standard education materials and tested on their confidence with their immunization decision
  Arms: Standard education only
Behavioral: Standard Education Plus OIDA — 50% of non-immunized personnel 4 weeks following start of campaign will be given standard education materials and tested on their confidence with their immunization decision
  Arms: Standard Education plus OIDA

SUMMARY:
The purpose of this study is to determine whether, among healthcare personnel who are undecided about whether to receive influenza vaccine, does use of the OIDA increase or decrease their confidence in their decision to be immunized? Furthermore, does the use of the OIDA affect the intent of the healthcare personnel to be immunized or not immunized?

DETAILED DESCRIPTION:
Influenza is one of the leading causes of acute respiratory infection and results in significant increases in average life-years lost, hospital lengths of stay and outpatient clinic visits, representing an enormous economic burden for many countries. Healthcare personnel are at particularly high risk of exposure to influenza as they are exposed in both the community and in the workplace. Influenza vaccination for healthcare personnel has been shown to reduce patient mortality in long-term care facilities as well as employee absenteeism and financial costs in acute care settings. The Canadian National Advisory Committee on Immunization (NACI) recommends that influenza immunization programs strive to immunize at least 90% of eligible recipients. In fact, NACI regards influenza immunization of healthcare personnel with direct patient care responsibilities as an essential component of the standard of care for the protection of patients. They consider the refusal of healthcare personnel without contraindications to receive influenza vaccine as a failure in their duty of care to patients. Despite national recommendations and proven effectiveness, influenza immunization coverage rates among healthcare personnel remain disappointingly low. In Canada, coverage rates among healthcare personnel range from 26-61% while in the US only 38% of healthcare personnel were immunized in 2002.

The decision to accept or refuse influenza vaccine each year may be a difficult one for many healthcare personnel. Decisional conflict, a term used to describe the difficulty experienced by an individual who simultaneously tends to both accept and reject a given course of action, occurs in many medical decisions where the best choice often differs depending on how individuals weigh the risks and benefits, and has been shown to contribute to poor vaccine uptake. In a review of literature from 1985 to 2004, it was found that healthcare personnel experience decisional conflict related to misperceptions about influenza, its risks, the role of healthcare personnel in its transmission to patients, and the importance and risks of vaccination.

Patient decision aids are tools that help people become involved in decision making by providing information about the options and outcomes, and clarifying personal values. They are designed to complement, rather than replace, counselling from a health practitioner. The use of decision aids has been shown to decrease decisional conflict and result in improved knowledge, more realistic expectations of benefit/risks and more active participation of individuals in decision-making. To date, no decision aids have been published that focus on influenza vaccination and none have been developed for healthcare personnel. Furthermore, the effect of a decision aid on the uptake of vaccine in healthcare personnel is unknown.

The peer-reviewed Ottawa Influenza Decision Aid (OIDA) was developed to respond to the aforementioned misconceptions and identify barriers of vaccine uptake in healthcare personnel. The OIDA presents evidence-based information and guides the individual through the decision-making process, including deliberation of personal values and beliefs.

ELIGIBILITY:
Inclusion Criteria:

For the purposes of this trial, the participating healthcare organizations will be required to:

1. Access a database of all healthcare personnel for whom influenza immunization is recommended
2. Collect real-time individual level immunization data about when healthcare personnel receive the vaccine
3. Generate a line-listing of all healthcare personnel for whom immunization status is not yet known at a pre-specified point in the campaign (at the end of the first four weeks of the campaign)
4. Contact the identified healthcare personnel in a manner approved by the healthcare organization, for example, by mail or e-mail, about participating in the trial
5. Ideally, have an institutional policy or high-level agreement that requires all healthcare personnel to provide evidence of their immunization status to occupational health.
6. Agree to work with the project team to boost the response rate, potentially by providing small tokens of appreciation to staff who complete the questionnaire or by promoting the study through regular communication channels (such as their internal network).

Exclusion Criteria:

Any organization not fitting above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Level of Confidence in Individual Healthcare Personnel in their Decision to be Immunized or not Against Influenza | 4 weeks after campaign start
  The level of confidence with which healthcare personnel reached a decision regarding immunization will be operationalized as a five-point ordinal scale with values ranging between 1 and 5.

SECONDARY OUTCOMES:
Do Healthcare Personnel Decide to be Immunized After Completing the OIDA? | 4 weeks after campaign start
  In keeping with the second objective of the trial, which is to measure the individual healthcare worker's decision to become immunized, the corresponding outcome measure is defined as a nominal variable registering the healthcare worker's self-reported course of action, to be used for estimating the rate of influenza immunization in each arm of the trial. In addition, the Occupational Health Department will provide information about the level of overall healthcare personnel immunization during running of the campaign after its first four weeks of operation.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E. McCarthy, MD, Principal Investigator — Ottawa Hospital Research Institute; Larry W Chambers, PhD(Epi), Principal Investigator — Bruyère Health Research Institute.
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Élisabeth Bruyère Research Institute, Ottawa, Ontario

REFERENCES:
- [Background] Lam PP, Chambers LW, MacDougall DM, McCarthy AE. Seasonal influenza vaccination campaigns for health care personnel: systematic review. CMAJ. 2010 Sep 7;182(12):E542-8. doi: 10.1503/cmaj.091304. Epub 2010 Jul 19. PMID 20643836